CLINICAL TRIAL: NCT00564486
Title: Phase 3 Randomized, Double-Blind Placebo-Controlled, Multicenter, Parallel-Group, Repeated-Dose Study of the Analgesic Efficacy & Safety of IV Acetaminophen Versus Placebo for the Treatment of Postop Pain
Brief Title: Analgesic Efficacy & Safety of Intravenous (IV) Acetaminophen Versus Placebo for the Treatment of Postop Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPI-APA-304
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Results first posted 2010-11-30 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Pain
Keywords: Abdominal Laparoscopic Surgery
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- IV Placebo 100 ml (Placebo Comparator): IV Placebo 100 ml dosed every every 6 hours for 24 hours (4 doses total).
  Interventions: Drug: IV Placebo
- IV Placebo 65 ml (Placebo Comparator): IV Placebo 65 ml dosed every every 4 hours for 24 hours (6 doses total).
  Interventions: Drug: IV Placebo
- IV Acetaminophen 1 gm (Experimental): IV Acetaminophen 1 gm dosed every every 6 hours for 24 hours (4 doses total).
  Interventions: Drug: IV Acetaminophen
- IV Acetaminophen 650 mg (Experimental): IV Acetaminophen 650 mg dosed every every 4 hours for 24 hours (6 doses total).
  Interventions: Drug: IV Acetaminophen

INTERVENTIONS:
Drug: IV Placebo — IV, every 6 hours for 24 hours (4 doses total)
  Other Names: placebo
  Arms: IV Placebo 100 ml
Drug: IV Placebo — IV, every 4 hours for 24 hours (6 doses total)
  Other Names: placebo
  Arms: IV Placebo 65 ml
Drug: IV Acetaminophen — IV, every 6 hours for 24 hours (4 doses total)
  Other Names: APAP; IV APAP
  Arms: IV Acetaminophen 1 gm
Drug: IV Acetaminophen — IV, every 4 hours for 24 hours (6 doses total)
  Other Names: APAP; IV APAP
  Arms: IV Acetaminophen 650 mg

SUMMARY:
This research study will look at the pain relieving ability and safety of using repeated doses of intravenous (into the vein [IV]) acetaminophen in the treatment of moderate postoperative pain after planned or elective abdominal laparoscopic surgery, such as a laparoscopic abdominal hysterectomy or laparoscopic cholecystectomy (removal of the gall bladder).

DETAILED DESCRIPTION:
To assess the analgesic efficacy of repeated doses of intravenous acetaminophen (IV APAP) versus Placebo in the treatment of moderate postoperative pain after abdominal laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Provide written Informed Consent prior to participation in the Study
* Is scheduled to undergo abdominal laparoscopic surgery under general anesthesia (laparoscopic bariatric procedures, including gastric bypass or gastric banding, laparoscopic exploratory procedures in which no visceral dissection is performed, and laparoscopic procedures with minimal visceral dissection, such as laparoscopic sterilization,are excluded)
* If Subject is a female of childbearing potential, have a negative pregnancy test within 21 days of surgery
* Be at least 18, but not more than 80 years of age
* Have a Body Mass Index (BMI) ≥ 19 and ≤ 40 lb/in2
* Have an American Society of Anesthesiologist (ASA) risk class of I, II, or III
* Have the ability to read and understand the Study procedures and the use of the pain scales and have the ability to communicate meaningfully with the Study Investigator and staff
* Be free of other physical, mental, or medical conditions which, in the opinion of the Investigator, makes Study participation inadvisable

Exclusion Criteria:

* Used opioids or tramadol daily for greater than 7 days prior to Study Medication administration (Subjects who, in the Investigator's opinion have or are developing opioid tolerance are to be excluded)
* Has been treated with Chapparal, Comfrey, Germander, Gin Bu Huan, Kava, Pennyroyal, Skullcap, St. John's Wort, or Valerian within 14 days prior to surgery
* Has significant medical disease(s), laboratory abnormalities or condition(s) that in the Investigator's judgment could compromise the Subject's welfare, ability to communicate with the Study staff, complete Study activities, or would otherwise contraindicate Study participation
* Has known hypersensitivity to opioids, acetaminophen, or the inactive ingredients (excipients) of the Study Medication
* Has known or suspected history of alcohol or drug abuse or dependence within the previous 2 years
* Has impaired liver function, e.g., aspartate aminotransferase (AST)/Alanine transaminase (ALT)/bilirubin greater than or equal to 3.0 times the upper limit of normal, active hepatic disease, evidence of clinically significant liver disease, or other condition (e.g., alcoholism, cirrhosis, or hepatitis) that may suggest the potential for an increased susceptibility to hepatic toxicity with Study Medication exposure
* Has been treated with monoamine oxidase inhibitors (MAOIs) within 7 days prior to surgery
* Has participated in another clinical Study (investigational or marketed product) within 30 days of surgery

Post Operative Exclusion Criteria

The Subject must not meet any of the following criteria prior to randomization to Study Medication:

* Had any other surgery than the planned laparoscopic surgery or had intra operative or post operative complications which in the view of the Investigator would make Study participation inadvisable
* Has taken non steroidal anti-inflammatory drugs (NSAIDs), steroids or MAOIs during the day after surgery. Exceptions: The use of low-dose aspirin, e.g, 81 mg/day, for cardioprophylaxis, and limited use of topical or inhaled steroids are acceptable.
* Had any neuraxial (spinal or epidural) opioid injected perioperatively
* Had a local anesthetic injection (including into surgical wound at closure) or continuous infusion by any route
* Had an epidural, regional, or percutaneous (intrawound) catheter with continuous local anesthetic infusion used for postoperative analgesic management
* Had a fever (greater than 38.6 ºC or 101.5 ºF) requiring treatment

Post Operative Day 1 Randomization Criterion On the morning of the first post operative day (POD1), the Subject must have a categorical pain intensity score at rest of moderate or severe and a score ≥ 40 mm and ≤ 70 mm at rest on a 100 mm Visual Analogue Scale (VAS)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Helen Keller Hospital, Sheffield, Alabama
  - Precision Trials, Phoenix, Arizona
  - Methodist Hospital, Arcadia, California
  - Glendale Adventist Medical Center, Glendale, California
  - Physicians Clinical Research Corporation, Laguna Hills, California
  - Huntington Memorial Hospital, Pasadena, California
  - Visions Clinical Research, Boynton Beach, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - G and G Research, Inc., Ft. Pierce, Florida
  - Advanced Surgery Associates at Mercy Hospital, Miami, Florida
  - University of Miami School of Medicine, Miami, Florida
  - William Beaumont Hospital (Royal Oak), Royal Oak, Michigan
  - William Beaumont Hospital (Troy), Royal Oak, Michigan
  - Cooper University Hospital, Camden, New Jersey
  - Staten Island University Hospital, Staten Island, New York
  - Memorial Herman/Memorial City Hospital, Houston, Texas
  - Texas Woman's Hospital, Houston, Texas

REFERENCES:
- [Derived] Wininger SJ, Miller H, Minkowitz HS, Royal MA, Ang RY, Breitmeyer JB, Singla NK. A randomized, double-blind, placebo-controlled, multicenter, repeat-dose study of two intravenous acetaminophen dosing regimens for the treatment of pain after abdominal laparoscopic surgery. Clin Ther. 2010 Dec;32(14):2348-69. doi: 10.1016/j.clinthera.2010.12.011. PMID 21353105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 sites across the US from 27 Nov 2007 to 12 September 2008.
Pre-assignment Details: On the morning of Post Operative Day 1, the subject was to have a pain intensity (PI) categorical score of moderate or severe and a visual analog scale (VAS) >= 40 mm, but <= 70 mm at rest on a 100 mm VAS.
Groups:
- Intravenous (IV) Placebo (100 ml): IV Placebo 100 ml dosed every every 6 hours for 24 hours (4 doses total).
- IV Placebo (65 ml): IV Placebo 65 ml dosed every every 4 hours for 24 hours (6 doses total).
Period: Overall Study
Arm/Group | Intravenous (IV) Placebo (100 ml) | IV Acetaminophen 1 gm | IV Acetaminophen 650 mg | IV Placebo (65 ml)
Started | 43 | 92 (One subject was randomized to receive 1 g IVAPAP but was administered 650 mg IV in error) | 42 (One subject randomized to receive 1 g IVAPAP but was administered 650 mg IV in error) | 67
Completed | 36 (Includes all subjects who returned to clinic for Day 7 visit.) | 91 (Includes all subjects who returned to clinic for Day 7 visit.) | 39 (Includes all subjects who returned to clinic for Day 7 visit.) | 60
Not Completed | 7 | 1 | 3 | 7
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 5
Not completed — Subject refused to have blood drawn | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- IV Placebo: All subjects randomized to receive IV Placebo 100 ml and IV placebo 65 ml groups combined
- IV Acetaminophen 1 gm: All subjects randomized to receive IV Acetaminophen 1 gm
- IV Acetaminophen 650 mg: All subjects randomized to receive IV Acetaminophen 650 mg
- Total: Total of all reporting groups
Arm/Group | IV Placebo | IV Acetaminophen 1 gm | IV Acetaminophen 650 mg | Total
Number analyzed (Participants) | 110 | 92 | 42 | 244
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 100 | 86 | 38 | 224
  >=65 years | 10 | 6 | 4 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 74 | 33 | 198
  Male | 19 | 18 | 9 | 46

OUTCOME MEASURES:

1. Primary Outcome: Sum Pain Intensity Difference - Baseline to 24 Hours (SPID24), 1 g IV Acetaminophen vs. Placebo (PI Was Measured at the Timepoints of T0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16, 18, 20, and 24 Hours.)
Description: Pain Intensity (PI) as measured by a 100 millimeter (mm) long Visual Analogue Scale (VAS) over 24 hours after treatment minus the Baseline VAS score. The 100 mm VAS was drawn on a pain ruler and labeled at its left end with '0 = No Pain' and with "100 = Worst Pain Imaginable' at its right end. Subjects placed a mark on the scale to represent their perceived pain. The score was the distance in mm from the left end of the VAS to the point where the subject's mark crossed the line. PI at baseline was compared to the PI at each timepoint and differences were summed over the 24 hour time period.
Time Frame: Baseline to 24 hrs
Population: All efficacy analyses were conducted using the modified intent-to-treat (mITT) population, defined as those subjects who received at least one complete infusion of study medication prior to requesting rescue medication.Worst Observation Carried Forward (WOCF) imputation was applied after first rescue medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- IV Placebo: mITT - IV Placebo 100 ml and IV placebo 65 ml groups combined
- IV Acetaminophen 1 gm: mITT - IV Acetaminophen 1 gm
Arm/Group | IV Placebo | IV Acetaminophen 1 gm
Number analyzed (Participants) | 108 | 92
Units on a scale | -45.2 (513.25) | -194.1 (593.62)

2. Secondary Outcome: Sum Pain Intensity Difference - Baseline to 24 Hours (SPID24), 650 mg IV Acetaminophen vs. Placebo (PI Was Measured at the Timepoints of T0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16, 18, 20, and 24 Hours.)
Description: Sum of Pain Intensity (PI) as measured by the 100 mm long Visual Analogue Scale (VAS) over 24 hours after treatment subtracting the Baseline VAS score.The 100 mm VAS was drawn on a pain ruler and labeled at it's left end with "0 = No Pain' and its right end with '100 = Worst Pain Imaginable.' Subjects placed a mark on the scale to represent their perceived pain. The score was the distance in mm from the left end of the VAS to the point where the subject's mark crossed the line. PI difference from baseline was calculated at each assessment over a 24 hour period.
Time Frame: Baseline to 24 hrs
Population: Included modified Intent To Treat group (mITT), defined as randomized subjects who received at least one complete infusion of study medication prior to receiving rescue medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- IV Acetaminophen 650 mg: mITT - IV Acetaminophen 650 mg
Arm/Group | IV Placebo | IV Acetaminophen 650 mg
Number analyzed (Participants) | 108 | 41
Units on a scale | -45.2 (513.25) | -323.1 (619.27)

3. Secondary Outcome: The Number of Subjects Reporting a Treatment Emergent Adverse Event
Description: Number of subjects who experienced at least one treatment emergent adverse event (TEAE).
  A TEAE is an adverse event that occurs on or after the first dose of study medication (T0).
Time Frame: First dose through 7 day follow up
Population: All analyses of safety were conducted on the safety population, which included those subjects who received any portion of a dose of study medication.
Measure: Number; unit: Subjects
Groups:
- IV Placebo: IV Placebo 100 ml and IV placebo 65 ml groups combined
- IV Acetaminophen 1000 mg: IV Acetaminophen 1000 mg every 6 hours for 24 hours
- IV Acetaminophen 650 mg: IV Acetaminophen 650 mg every 4 hours for 24 hours
Arm/Group | IV Placebo | IV Acetaminophen 1000 mg | IV Acetaminophen 650 mg
Number analyzed (Participants) | 110 | 91 | 43
Subjects | 68 | 65 | 28

4. Secondary Outcome: The Number of Subjects Reporting a Treatment Emergent Serious Adverse Event
Description: The number of subjects who reported at least one treatment emergent SAE during the study.
  A Serious Adverse Event is defined as any untoward medical occurrence at any dose of blinded study medication that:
  * results in death
  * is life-threatening
  * requires inpatient hospitalization or causes prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
  * is an important medical event
Time Frame: First dose to 30 days after last dose of study medication.
Population: All analyses were conducted on the safety population, which included those subjects who received any portion of a dose of study medication.
Measure: Number; unit: Subjects
Groups:
- IV Acetaminophen 1 gm: IV Acetaminophen 1 gm every 6 hours for 24 hours (4 doses total)
- IV Acetaminophen 650 mg: IV Acetaminophen 650 mg every 4 hours for 24 hours (6 doses total)
Arm/Group | IV Placebo | IV Acetaminophen 1 gm | IV Acetaminophen 650 mg
Number analyzed (Participants) | 110 | 91 | 43
Subjects | 2 | 1 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from T0 (on or after start of study drug) to Day 7 after surgery. Serious Adverse Events were collected from T0 to 30 days after the last dose of study medication.
Arm/Group | Intravenous (IV) Placebo (100 ml) | IV Acetaminophen 1 gm | IV Acetaminophen 650 mg | IV Placebo (65 ml)
Serious Adverse Events (participants affected / at risk) | 0/43 | 1/91 | 3/43 | 2/67
Other Adverse Events (participants affected / at risk) | 12/43 | 42/91 | 16/43 | 27/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous (IV) Placebo (100 ml) (N=43) | IV Acetaminophen 1 gm (N=91) | IV Acetaminophen 650 mg (N=43) | IV Placebo (65 ml) (N=67)
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous (IV) Placebo (100 ml) (N=43) | IV Acetaminophen 1 gm (N=91) | IV Acetaminophen 650 mg (N=43) | IV Placebo (65 ml) (N=67)
Constipation (Gastrointestinal disorders) | 7 | 16 | 5 | 11
Flatulence (Gastrointestinal disorders) | 4 | 14 | 4 | 6
Nausea (Gastrointestinal disorders) | 3 | 16 | 4 | 9
Vomiting (Gastrointestinal disorders) | 0 | 7 | 4 | 2
Headache (Nervous system disorders) | 4 | 12 | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 0 | 5
Infusion site pain (General disorders) | 0 | 5 | 1 | 1
Pyrexia (General disorders) | 5 | 2 | 0 | 2
Incision site pain (Injury, poisoning and procedural complications) | 0 | 5 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 6
Insomnia (Psychiatric disorders) | 1 | 2 | 3 | 4
Dypsnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0

LIMITATIONS AND CAVEATS:
One subject was randomized to receive IV APAP 1 g, but was administered IV APAP 650 mg. The subject was included in 1g IV APAP group for efficacy purposes and included in IV APAP 650 mg safety group for AE purposes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution or Investigator may publish the results of the study (without raw data, detailed patient Case Report Forms, or patient identification) only after such cooperative publication, or 18 months after Cadence's final evaluation of all study data from all sites, whichever occurs first. At least 60 days prior to submission, or prior to any public presentation, a copy of the abstract, manuscript or presentation will be provided to Cadence who will have 60 days to respond with comments.